CLINICAL TRIAL: NCT01840618
Title: Effect of Obstructive Sleep Apnea Syndrome on Insulin Sensitivity and Cardiovascular Risk in PCOS Adolescents
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 11-09-336E
Record Dates: First submitted 2012-07-12; First posted 2013-04-26 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Obstructive Sleep Apnea Syndrome; Polycystic Ovary Syndrome; Sleep Apnea
Keywords: insulin function; sleep apnea; girls; PCOS; insulin action
MeSH Terms: conditions — Sleep Apnea, Obstructive; Polycystic Ovary Syndrome; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Obese PCOS and sleep apnea: BMI >95%ile AND Polysomnography with AHI >2.5
  Will initiate Nasal Continuous positive airway pressure (CPAP)
  Interventions: Device: Nasal Continuous positive airway pressure (CPAP)
- Obese PCOS without sleep apnea: BMI >95%ile AND Polysomnography with AHI <2.5
- Normal weight Controls: BMI <85%ile AND regular menses
- Lean PCOS and sleep apnea: BMI <85%ile AND Polysomnography with AHI >2.5
  Will initiate Nasal Continuous positive airway pressure (CPAP)
  Interventions: Device: Nasal Continuous positive airway pressure (CPAP)
- Lean PCOS without sleep apnea: BMI <85%ile AND Polysomnography with AHI <2.5

INTERVENTIONS:
Device: Nasal Continuous positive airway pressure (CPAP) — We will initiate treatment of OSA with CPAP for 3 months in PCOS adolescents with moderate to severe OSA. Compliance will be defined as the average number of hours for which CPAP was used per night over the 12-wk treatment period. Adherence with CPAP will be defined as CPAP use ≥4 hours daily. The primary outcome variable will be insulin sensitivity measured as change in GIR. Changes in cardio metabolic variables after CPAP treatment will be expressed as a percentage of the corresponding baseline values.
  Groups: Lean PCOS and sleep apnea; Obese PCOS and sleep apnea

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common disease caused by hormonal imbalance and is also associated with overweight and obesity. It affects 5-10% of adolescent girls and women capable of having children. Polycystic ovary syndrome is associated with missed menstrual periods, hormonal imbalance, being overweight, and with a form of diabetes. Girls with polycystic ovary syndrome may have a breathing problem known as "sleep apnea." Sleep apnea may cause a person to stop breathing for short periods of time while sleeping. People with polycystic ovary syndrome are thirty times more likely to develop sleep apnea than those who do not have PCOS. If sleep apnea is not treated, it may lead to daytime sleepiness, poor school performance, high blood pressure, heart disease and diabetes. The purpose of this study is to understand how insulin function is affected in presence of sleep apnea in girls with polycystic ovary syndrome between 13-21 years of age as compared to girls with PCOS without sleep apnea. Insulin is one of the hormones made in your body to convert food into energy. In people with increase weight body cannot use insulin properly. The investigators also want to see if insulin action is also affected by sleep apnea.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Ages 13-21
* PCOS
* BMI >95%ile (Obese group) or <85%ile (Lean group)
* Controls: ages 18-21, regular menses, BMI <85%ile

Exclusion Criteria:

* Breastfeeding.
* Pregnant.
* Use of any steroid preparations (including hormonal contraception), medications known to alter insulin secretion and/or action within 3 month (including Metformin)

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Girls with PCOS, with and without sleep apnea. Ages 13-21.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to understand how insulin function is affected and how endothelial function as a surrogate marker for cardiovascular risk is affected in presence of sleep apnea as compared to girls (13-21 yrs) with PCOS without sleep apnea | baseline to two years
  Obese adolescents with PCOS will be assessed for presence or absence of Obstructive Sleep Apnea (OSA) at baseline. Obese PCOS with OSA will be compared with obese PCOS with out OSA for difference in Glucose Infusion Rate (GIR) as a measure of insulin resistance and for Reactive Hyperemia Peripheral Arterial Tonometry (RHPAT) score

SECONDARY OUTCOMES:
We also want to see if there is any change in the levels of adipocytokines (Leptin, adiponectin, C Reactive Protein (CRP), Tumor Necrosis Factor (TNF) alpha, Free fatty acids) because of sleep apnea in obese PCOS adolescents. | baseline to two years
  Obese adolescents with PCOS will be assessed for presence or absence of Obstructive Sleep Apnea (OSA) at baseline. Obese PCOS with OSA will be compared with obese PCOS with out OSA for increase in the levels of leptin, CRP, TNF alpha, free fatty acids and the reduction in the levels of adiponectin compared to Non OSA adolescents with PCOS.

OTHER OUTCOMES:
The purpose of this study is to to determine the role that PCOS plays in insulin resistance in non-obese adolescents by comparing insulin resistance in adolescent girls ages 13-21 with lean PCOS to normal weight adolescents ages 18-21 without PCOS. | baseline to two years
  Insulin sensitivity will be compared in adolescents with non-obese PCOS (BMI ≤85%) to non-obese adolescents (BMI ≤85%) without PCOS

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Underland, MD, Principal Investigator — Montefiore Medical Center, Albert Einstein
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States